CLINICAL TRIAL: NCT05490277
Title: Vibrotactile Coordinated Reset for the Treatment of Chronic Stroke
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Peter Tass, MD, PhD, Protocol Director, Stanford University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 65197
Record Dates: First submitted 2022-08-02; First posted 2022-08-05 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2024-08

CONDITIONS: Chronic Stroke

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Active Vibrotactile Coordinated Reset (vCR) (Active Comparator): Vibrotactile Coordinated Reset delivers vibratory stimulation to the fingertips of each hand. A specific pattern of vibration to each fingertip is delivered which theoretically disrupts abnormal synchrony in the brain.
  Interventions: Device: Active Vibrotactile coordinated reset
- Sham Vibrotactile Coordinated Reset (vCR) (Sham Comparator): Vibrotactile Coordinated Reset delivers vibratory stimulation to the fingertips of each hand. An inactive pattern of vibration to each fingertip is delivered which theoretically will not have the effects of active vCR.
  Interventions: Device: Sham vibrotactile coordinated reset

INTERVENTIONS:
Device: Active Vibrotactile coordinated reset — Participants will receive active vibrotactile coordinated reset (vCR) which sends gentle vibrations to the fingertips at a specific pattern. The purpose of the intervention is to test the efficacy of active vCR in comparison to sham vCR.
  Arms: Active Vibrotactile Coordinated Reset (vCR)
Device: Sham vibrotactile coordinated reset — Participants will receive sham vibrotactile coordinated reset (vCR) which sends gentle vibrations to the fingertips at a specific pattern. The purpose of the intervention is to test the efficacy of active vCR in comparison to sham vCR.
  Arms: Sham Vibrotactile Coordinated Reset (vCR)

SUMMARY:
The purpose of our study is to evaluate Vibrotactile Coordinated Reset stimulation (vCR) and its effects on motor ability within stroke patients. vCR will be administered with a device called the Vibrotactile (VT) Brain Glove. vCR is expected to provide patients with a non-invasive therapy to aid in recovery from a stroke. This study will include a dedicated sham arm that will aid in understanding true treatment effects from vCR.

ELIGIBILITY:
Inclusion Criteria:

1. Age at the time of enrollment: 18-80 years
2. Diagnosis of ischemic or hemorrhagic stroke
3. Disease period of more than 6 months
4. Mini Mental State Examination of at least 24 points
5. No medications that affect balance
6. Motor deficit
7. Use of Motricity Arm and Leg index to include impaired individuals with some functioning
8. Modified Rankin Scale for Neurologic Disability: Scores 3 or 4

Exclusion Criteria:

1. Any significant psychiatric problems, including acute confusional state (delirium), ongoing psychosis, or clinically significant depression
2. Any current drug or alcohol abuse
3. History of recurrent or unprovoked seizures
4. Any neurological disorder treatments that involve intracranial surgery or device implantation
5. Participation in another drug, device or biologic trial concurrently or within the preceding days
6. Pregnancy, breastfeeding or wanting to become pregnant during the trial
7. History or presence of other major neurological or orthopedic diseases other than stroke that limits motor functioning or cognitive ability
8. More than 5 degrees of contracture at shoulder, elbow, wrist, finger, hip, knee, or ankle
9. Botox, baclofen or any other treatment for spasticity except for bracing or splinting within the previous 3 months
10. Must be able to communicate with staff
11. Severe sensory abnormalities of the fingers such as vibratory urticaria

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2028-11-15 (Estimated); Study Completion 2028-11-15 (Estimated)

PRIMARY OUTCOMES:
Fugl Meyer Assessment of Motor Recovery after Stroke change from baseline, 3 months, 4 months, 7months and 8 months | This clinical assessment will be done at baseline visit, three month visit, four month visit, seven month visit and eight month visit
  The Fugl-Meyer Assessment (FMA) is a stroke-specific, performance-based impairment index. It is designed to assess motor functioning, balance, sensation and joint functioning in patients with post-stroke hemiplegia. It is applied clinically and in research to determine disease severity, describe motor recovery, and to plan and assess treatment. The scale is comprised of five domains and there are 155 items in total. Scoring is based on direct observation of performance. Scale items are scored on the basis of ability to complete the item using a 3-point ordinal scale where 0=cannot perform, 1=performs partially and 2=performs fully. The total possible scale score is 226.
Neuro Quality of Life Upper Extremity Short Form test change from baseline, 3 months, 4 months, 7months and 8 months | This clinical assessment will be done at baseline visit, three month visit, four month visit, seven month visit and eight month visit
  The Neuro quality of life upper extremity short form test measures the functionality of upper extremities. This is a self-report questionnaire that has a Likert scale from 1 to 5, with 5 indicating no difficulties and 1 indicating unable to do. Total possible points are out of 40, with a higher score indicating better upper extremity abilities.

SECONDARY OUTCOMES:
Barthel Index for Activities of Daily Living change from baseline, 3 months, 4 months, 7months and 8 months | This clinical assessment will be done at baseline visit, three month visit, four month visit, seven month visit and eight month visit
  The Barthel Index (BI) measures the extent to which somebody can function independently and has mobility in their activities of daily living (ADL) i.e. feeding, bathing, grooming, dressing, bowel control, bladder control, toileting, chair transfer, ambulation and stair climbing. Functional categories may be scored from 0 to 1, 0 to 2, or 0 to 3, depending on the item. Total scores range from 0 to 20, with lower scores indicating increased disability
Action Research Arm Test change from baseline, 3 months, 4 months, 7months and 8 months | This clinical assessment will be done at baseline visit, three month visit, four month visit, seven month visit and eight month visit
  The Action Research Arm Test (ARAT) is a 19 item observational measure used by physical therapists and other health care professionals to assess upper extremity performance (coordination, dexterity and functioning) in stroke recovery, brain injury and multiple sclerosis populations.Items comprising the ARAT are categorized into four subscales (grasp, grip, pinch and gross movement). Task performance is rated on a 4-point scale, ranging from 0 (no movement) to 3 (movement performed normally). Scores on the ARAT may range from 0-57 points, with a maximum score of 57 points indicating better performance.
Timed Up and Go test change from baseline, 3 months, 4 months, 7months and 8 months | This clinical assessment will be done at baseline visit, three month visit, four month visit, seven month visit and eight month visit
  This test is a measure walking ability with correlates to balance and fall risk. The patient is timed using a stopwatch and the patient is instructed to walk as quickly as possible for 3 meters. The test is scored as such: ≤ 10 seconds = normal ≤ 20 seconds = good mobility, can go out alone, mobile without gait aid ≤ 30 seconds = problems, cannot go outside alone, requires gait aid * A score of ≥ 14 seconds has been shown to indicate high risk of falls
Neuro Quality of Life Lower Extremity Short Form test change from baseline, 3 months, 4 months, 7months and 8 months | This clinical assessment will be done at baseline visit, three month visit, four month visit, seven month visit and eight month visit
  The Neuro quality of life lower extremity short form test measures the functionality of upper extremities. This is a self-report questionnaire that has a Likert scale from 1 to 5, with 5 indicating no difficulties and 1 indicating unable to do. Total possible points are out of 40, with a higher score indicating better lower extremity abilities.
Sensorimotor reaction time task | This clinical assessment will be done at baseline visit, three month visit, four month visit, seven month visit and eight month visit
  Patients receive vibratory stimuli on a finger and indicate when stimuli are felt by pressing a button.
Vibratory temporal discrimination task | This clinical assessment will be done at baseline visit, three month visit, four month visit, seven month visit and eight month visit
  Patients receive vibratory stimuli on two fingers either simultaneously or at different times and indicate the perceived timing by pressing a button.

CONTACTS AND LOCATIONS:
Overall Officials: Peter A Tass, MD, PhD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: Undecided
Individual participant data is deidentified and may be shared with other researchers upon request